CLINICAL TRIAL: NCT00683930
Title: A Prospective, Randomised, Double-blind, Placebo-controlled, Parallel Group, Mult-center, 52-week Trial to Assess the Efficacy and Safety of Adjunct Mycophenolate Mofetil (MMF) to Achieve Remission With Reduced Corticosteroid in Subjects With Pemphigus Vulgaris
Brief Title: A Study to Assess the Effect of CellCept (Mycophenolate Mofetil) and Reduced Corticosteroids in Patients With Active Pemphigus Vulgaris (PV)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Aspreva Pharmaceuticals (Industry)
Responsible Party: Disclosures Group, Hoffmann-La Roche
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WX17796; NCT00140127 (obsolete NCT alias)
Record Dates: First submitted 2008-05-19; First posted 2008-05-26 (Estimated); Results first posted 2011-06-22 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-05

CONDITIONS: Pemphigus Vulgaris (PV)
MeSH Terms: conditions — Pemphigus | interventions — Mycophenolic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Mycophenolate Mofetil (MMF) 2 g/Day (Experimental): Mycophenolate mofetil 500 mg tablets; 4 tablets twice daily for 52 weeks
  Interventions: Drug: Mycophenolate Mofetil 2 g/Day
- Mycophenolate Mofetil (MMF) 3 g/Day (Experimental): Mycophenolate mofetil 500 mg tablets; 6 tablets twice daily for 52 weeks
  Interventions: Drug: Mycophenolate Mofetil (MMF) 3 g/Day
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mycophenolate Mofetil 2 g/Day — Mycophenolate mofetil 500 mg tablets; 4 tablets twice daily for 52 weeks
  Arms: Mycophenolate Mofetil (MMF) 2 g/Day
Drug: Mycophenolate Mofetil (MMF) 3 g/Day — Mycophenolate mofetil 500 mg tablets; 6 tablets twice daily for 52 weeks
  Arms: Mycophenolate Mofetil (MMF) 3 g/Day
Drug: Placebo — Placebo for MMF 2 g/day group: 4 tablets orally twice daily for 52 weeks; placebo for MMF 3 g/day group: 6 tablets orally twice daily for 52 weeks
  Arms: Placebo

SUMMARY:
This study was designed to assess the efficacy and safety of CellCept (1 g or 1.5 g orally twice daily for 52 weeks) in patients with pemphigus vulgaris receiving prednisone or other corticosteroids. During the study, patients had their corticosteroid dose gradually reduced if they responded to treatment. The anticipated time on study treatment was 12 months, and the target sample size was <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18 to 70 years of age
* Diagnosis of mild to moderate pemphigus vulgaris within the past 12 months, requiring high dose corticosteroids

Exclusion Criteria:

* Female patients who are pregnant, breastfeeding, or lactating
* Regularly scheduled plasma exchange (PE) or intravenous immunoglobulin (IVIG) treatment, or PE or IVIG treatment within 8 weeks prior to randomization
* CellCept or other immunosuppressive therapy, except corticosteroids, exceeding 2 weeks total duration and within 8 weeks prior to randomization
* Use of PV therapies other than those noted above, within 4 weeks prior to randomization
* Use of topical corticosteroids within 2 weeks prior to randomization

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2004-05; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (25):
- United States (5):
  - Los Angeles, California
  - Atlanta, Georgia
  - Baltimore, Maryland
  - St Louis, Missouri
  - New York, New York
- Canada (2):
  - Toronto, Ontario
  - Montreal, Quebec
- Germany (6):
  - Cologne
  - Frankfurt am Main
  - Heidelberg
  - Mainz
  - Münster
  - Ulm
- Israel (2):
  - Haifa
  - Petah Tikva
- Zurich, Switzerland
- Turkey (Türkiye) (2):
  - Ankara
  - Istanbul
- Ukraine (5):
  - Crimea
  - Donetsk
  - Kiev
  - Lugnansk
  - Uzhhorod
- United Kingdom (2):
  - Leicester
  - London

REFERENCES:
- [Derived] Beissert S, Mimouni D, Kanwar AJ, Solomons N, Kalia V, Anhalt GJ. Treating pemphigus vulgaris with prednisone and mycophenolate mofetil: a multicenter, randomized, placebo-controlled trial. J Invest Dermatol. 2010 Aug;130(8):2041-8. doi: 10.1038/jid.2010.91. Epub 2010 Apr 22. PMID 20410913

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo for Mycophenolate Mofetil (MMF) 2 g/day group: 4 tablets orally twice daily for 52 weeks; placebo for MMF 3 g/day group: 6 tablets orally twice daily for 52 weeks
- MMF 2 g/Day: Mycophenolate mofetil (MMF) 500 mg tablets; 4 tablets twice daily for 52 weeks
- MMF 3 g/Day: Mycophenolate mofetil (MMF) 500 mg tablets; 6 tablets twice daily for 52 weeks
Period: Overall Study
Arm/Group | Placebo | MMF 2 g/Day | MMF 3 g/Day
Started | 36 (One subject not included: no study drug dispensed.) | 21 (One subject not included: no study drug dispensed.) | 37
Completed | 29 | 18 | 28
Not Completed | 7 | 3 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | MMF 2 g/Day | MMF 3 g/Day | Total
Number analyzed (Participants) | 36 | 21 | 37 | 94
Age Continuous [Mean (Standard Deviation); unit: years] — Intent-to-treat population
  years | 45.8 (12.18) | 41.0 (15.59) | 44.8 (13.47) | 44.33 (13.45)
Sex: Female, Male [Count of Participants; unit: Participants] — Intent-to-treat population
  Participants
    Female | 24 | 14 | 18 | 56
    Male | 12 | 7 | 19 | 38

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Achieving Responder Status at Week 52
Description: The proportion of subjects achieving responder status (defined as no new persistent lesions and prednisone dose of not more than 10 mg/day from Week 48 until study termination at Week 52) in the two active treatment groups combined (2 g/day and 3 g/day mycophenolate mofetil) compared with the placebo group
Time Frame: 52 weeks
Population: Intent-to-treat population. Analysis population (AP): Placebo = 36; MMF 2 g/day or 3 g/day = 58.
Measure: Number; unit: Percentage of Participants
Groups:
- MMF 2 g/Day and MMF 3 g/Day Groups Combined: MMF 2 g/day group: 500 mg tablets, 4 tablets twice daily for 52 weeks MMF 3 g/day group: 500 mg tablets, 6 tablets twice daily for 52 weeks
Arm/Group | Placebo | MMF 2 g/Day and MMF 3 g/Day Groups Combined
Number analyzed (Participants) | 36 | 58
Percentage of Participants | 63.9 | 69.0
Statistical Analysis 1: Comparison: Placebo vs MMF 2 g/Day and MMF 3 g/Day Groups Combined; Test type: Superiority or Other; p = 0.6558, Fisher Exact; Alpha = 0.025; Treatment difference in response rate = 5.1, 97.5% CI [-17.4 to 27.6]

2. Secondary Outcome: Time to Initial Response
Description: Time to initial response defined as the time that the subject first demonstrated responder status (defined as no new persistent lesions and prednisone dose of not more than 10 mg/day from Week 48 until study termination at Week 52)
Time Frame: up to 52 weeks
Population: Intent-to-treat population. Analysis population (AP): Placebo = 36, subjects censored = 7; MMF 2 g/day or 3 g/day = 58, subjects censored = 10.
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Placebo | MMF 2 g/Day and MMF 3 g/Day Groups Combined
Number analyzed (Participants) | 36 | 58
Weeks | 31.3 [25.0 to 36.4] | 24.1 [20.3 to 32.4]

3. Secondary Outcome: Time to Sustained Response
Description: Time to sustained response is defined as the week the subject first demonstrates both of the conditions of responder status provided the conditions are maintained through to study termination at Week 52. If a subject does not have a sustained response, time to sustained response is censored on the last day of the study.
Time Frame: up to 52 weeks
Population: Intent-to-treat population. Analysis population (AP): Placebo = 36, subjects censored = 20; MMF 2 g/day or 3 g/day = 58, subjects censored = 23.
Measure: Median (Full Range); unit: Weeks
Arm/Group | Placebo | MMF 2 g/Day and MMF 3 g/Day Groups Combined
Number analyzed (Participants) | 16 | 35
Weeks | 46.0 [29.7 to NA] — Data not available. Median, Q1, and Q3 are calculated from Kaplan-Meier estimates. | 32.1 [20.6 to NA] — Data not available. Median, Q1, and Q3 are calculated from Kaplan-Meier estimates.

4. Secondary Outcome: Duration of Prednisone Maintenance Dosing
Description: The duration of prednisone maintenance dosing was defined as the number of days that subjects maintained a prednisone dose of not more than 10 mg/day in the absence of new persistent lesions.
Time Frame: 52 weeks
Population: Intent-to-treat population. Analysis population (AP): Placebo = 36; MMF 2 g/day = 21; MMF 3 g/day = 37; MMF Groups Combined (2 g/day or 3 g/day) = 58.
Measure: Median (Inter-Quartile Range); unit: Days
Groups:
- Mycophenolate Mofetil 2 g/Day: MMF 500 mg tablets; 4 tablets twice daily for 52 weeks
- Mycophenolate Mofetil 3 g/Day: MMF 500 mg tablets; 6 tablets twice daily for 52 weeks
Arm/Group | Placebo | MMF 2 g/Day and MMF 3 g/Day Groups Combined | Mycophenolate Mofetil 2 g/Day | Mycophenolate Mofetil 3 g/Day
Number analyzed (Participants) | 36 | 58 | 21 | 37
Days | 136.5 [60.0 to 191.0] | 186.0 [79.0 to 244.0] | 185.0 [109.0 to 246.0] | 187.0 [75.0 to 225.0]

ADVERSE EVENTS:
Time Frame: AEs were monitored throughout the course of the study. Further follow-up was made at approximately 24 weeks (±7 days) after the Week 52 visit to record any AEs that occurred during the follow-up period.
Description: Safety analysis population. Note one patient from both the placebo group and MMF 2g/day group were excluded from the safety population as no study drug was dispensed.
Arm/Group | Placebo | MMF 2 g/Day | MMF 3 g/Day
Serious Adverse Events (participants affected / at risk) | 4/36 | 1/21 | 3/37
Other Adverse Events (participants affected / at risk) | 31/36 | 20/21 | 32/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=36) | MMF 2 g/Day (N=21) | MMF 3 g/Day (N=37)
Food Poisoning (Gastrointestinal disorders) | 1 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 1 | 0
Pemphigus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Cardiovascular Insufficiency (Vascular disorders) | 1 | 0 | 0
Duodenal Ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Varicella (Infections and infestations) | 0 | 0 | 1
Cataract (Eye disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=36) | MMF 2 g/Day (N=21) | MMF 3 g/Day (N=37)
Nasopharyngitis (Infections and infestations) | 0 | 4 | 3
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 1 | 5
Rhinitis (Infections and infestations) | 0 | 0 | 2
Laryngitis (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0 | 1
Oral Candidiasis (Infections and infestations) | 2 | 1 | 9
Candidiasis (Infections and infestations) | 2 | 1 | 1
Skin Candida (Infections and infestations) | 1 | 0 | 0
Skin Infection (Infections and infestations) | 1 | 2 | 1
Furuncle (Infections and infestations) | 0 | 0 | 2
Paronychia (Infections and infestations) | 0 | 0 | 1
Pyoderma (Infections and infestations) | 0 | 1 | 0
Subcutaneous Abscess (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 1
Bronchitis Acute (Infections and infestations) | 0 | 0 | 2
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0
Pneumonia Primary Atypical (Infections and infestations) | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 2 | 0 | 4
Cystitis (Infections and infestations) | 0 | 0 | 2
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Urethritis (Infections and infestations) | 1 | 0 | 0
Herpes Simplex (Infections and infestations) | 1 | 2 | 2
Herpetic Gingivostomatitis (Infections and infestations) | 0 | 0 | 2
Herpes Zoster (Infections and infestations) | 1 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 2
Bacteriuria (Infections and infestations) | 0 | 0 | 1
Bacterial Infection (Infections and infestations) | 1 | 0 | 0
Tinea Versicolour (Infections and infestations) | 0 | 1 | 2
Body Tinea (Infections and infestations) | 2 | 0 | 1
Viral Infection (Infections and infestations) | 0 | 0 | 2
Bronchitis Viral (Infections and infestations) | 0 | 0 | 1
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 1
Dysentery (Infections and infestations) | 1 | 0 | 0
Tooth Abscess (Infections and infestations) | 1 | 1 | 0
Fungal Skin Infection (Infections and infestations) | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 1
Molluscum Contagiosum (Infections and infestations) | 0 | 1 | 0
Anogenital Warts (Infections and infestations) | 1 | 0 | 0
Pemphigus (Skin and subcutaneous tissue disorders) | 12 | 7 | 10
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 4
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 1
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 1 | 1
Alopecia Effluvium (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Heat Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Swelling Face (Skin and subcutaneous tissue disorders) | 3 | 1 | 1
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Purpura Senile (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 4
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1
Constipation (Gastrointestinal disorders) | 2 | 2 | 3
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 3
Abdominal Pain (Gastrointestinal disorders) | 3 | 0 | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 0 | 2
Frequent Bowel Movements (Gastrointestinal disorders) | 0 | 1 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 1
Lip Ulceration (Gastrointestinal disorders) | 0 | 1 | 0
Oral Soft Tissue Disorder (Gastrointestinal disorders) | 1 | 0 | 0
Aphthous Stomatitis (Gastrointestinal disorders) | 1 | 1 | 0
Mouth Ulceration (Gastrointestinal disorders) | 1 | 0 | 1
Oral Mucosa Erosion (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Rectal Tenesmus (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 1
Abdominal Distension (Gastrointestinal disorders) | 1 | 0 | 1
Flatulence (Gastrointestinal disorders) | 2 | 0 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0
Stomach Discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Dry Mouth (Gastrointestinal disorders) | 0 | 1 | 0
Oral Pain (Gastrointestinal disorders) | 0 | 0 | 1
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 0
Oral Discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Salivary Hypersecretion (Gastrointestinal disorders) | 0 | 0 | 1
Anal Fissure (Gastrointestinal disorders) | 1 | 0 | 0
Loose Tooth (Gastrointestinal disorders) | 1 | 0 | 0
Gingivitis (Gastrointestinal disorders) | 2 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 3 | 4 | 3
Fatigue (General disorders) | 0 | 1 | 2
Asthenia (General disorders) | 1 | 0 | 2
Pain (General disorders) | 0 | 1 | 2
Chest Pain (General disorders) | 0 | 0 | 1
Irritability (General disorders) | 0 | 1 | 1
Influenza Like Illness (General disorders) | 0 | 0 | 1
Chest Discomfort (General disorders) | 1 | 0 | 0
Oedema Peripheral (General disorders) | 0 | 1 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Sensation of Heaviness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 2
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Muscle Twitching (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myopathy Steroid (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle Rigidity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 6
Dysgeusia (Nervous system disorders) | 0 | 2 | 2
Lethargy (Nervous system disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1
Migraine With Aura (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0
Post Herpetic Neuralgia (Nervous system disorders) | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1
Dyskinesia (Nervous system disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 3
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchial Hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2
Arthropod Bite (Injury, poisoning and procedural complications) | 1 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Arthropod Sting (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ear Abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Joint Sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Amenorrhoea (Reproductive system and breast disorders) | 0 | 2 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1
Polymenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0
Erectile Dysfunction (Reproductive system and breast disorders) | 0 | 0 | 1
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Perineal Pain (Reproductive system and breast disorders) | 0 | 0 | 1
Vaginal Erosion (Reproductive system and breast disorders) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 3 | 1 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 2
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocythaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 1 | 1
Vision Blurred (Eye disorders) | 0 | 1 | 0
Visual Disturbance (Eye disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 1 | 0
Glaucoma (Eye disorders) | 0 | 1 | 0
Lacrimation Increased (Eye disorders) | 0 | 1 | 0
Abnormal Sensation in Eye (Eye disorders) | 1 | 0 | 0
Weight Increased (Investigations) | 1 | 0 | 3
Weight Decreased (Investigations) | 0 | 0 | 1
Blood Glucose Increased (Investigations) | 0 | 1 | 0
Electrocardiogram ST-T Change (Investigations) | 0 | 0 | 1
Culture Urine Positive (Investigations) | 0 | 0 | 1
Sputum Culture Positive (Investigations) | 0 | 0 | 1
Intraocular Pressure Increased (Investigations) | 1 | 0 | 0
White Blood Cells Urine (Investigations) | 1 | 0 | 0
Hypertension (Vascular disorders) | 4 | 3 | 3
Venous Thrombosis (Vascular disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 2
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 1 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 1
Libido Decreased (Psychiatric disorders) | 0 | 1 | 0
Sleep Disorder (Psychiatric disorders) | 1 | 1 | 0
Nervousness (Psychiatric disorders) | 1 | 0 | 0
Depressed Mood (Psychiatric disorders) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 2
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 1
Cushingoid (Endocrine disorders) | 0 | 0 | 2
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 1
Allergy to Arthropod Bite (Immune system disorders) | 1 | 0 | 1
Central Obesity (Metabolism and nutrition disorders) | 0 | 0 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Iron Deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.